CLINICAL TRIAL: NCT06322056
Title: Exploring Approaches With Lower Targets of Blood Pressure and Lipid for Improving Renal Outcome in Advanced Chronic Kidney Disease
Acronym: EXCELSIOR-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1654
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases; Hypertension; Dyslipidemias
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intensive SBP control and Intensive LDL-C control (Active Comparator): Targeting SBP <120 mmHg and targeting LDL-C <70 mg/dL
  Interventions: Drug: Intensive control of SBP and intensive control of LDL-C
- Intensive SBP control and Standard LDL-C control (Active Comparator): Targeting SBP <120 mmHg and targeting LDL-C <100 mg/dL
  Interventions: Drug: Intensive control of SBP and standard control of LDL-C
- Standard SBP control and Intensive LDL-C control (Active Comparator): Targeting SBP <140 mmHg and targeting LDL-C <70 mg/dL
  Interventions: Drug: Standard control of SBP and intensive control of LDL-C
- Standard SBP control and Standard LDL-C control (Active Comparator): Targeting SBP <140 mmHg and targeting LDL-C <100 mg/dL
  Interventions: Drug: Standard control of SBP and standard control of LDL-C

INTERVENTIONS:
Drug: Intensive control of SBP and intensive control of LDL-C — Eligible participants would be assigned to a SBP target of less than 120 mmHg and a LDL-C target of less than 70 mg/dL.
  Arms: Intensive SBP control and Intensive LDL-C control
Drug: Intensive control of SBP and standard control of LDL-C — Eligible participants would be assigned to a SBP target of less than 120 mmHg and a LDL-C target of less than 100 mg/dL.
  Arms: Intensive SBP control and Standard LDL-C control
Drug: Standard control of SBP and intensive control of LDL-C — Eligible participants would be assigned to a SBP target of less than 140 mmHg and a LDL-C target of less than 70 mg/dL.
  Arms: Standard SBP control and Intensive LDL-C control
Drug: Standard control of SBP and standard control of LDL-C — Eligible participants would be assigned to a SBP target of less than 140 mmHg and a LDL-C target of less than 100 mg/dL.
  Arms: Standard SBP control and Standard LDL-C control

SUMMARY:
The purpose of this study is to prevent kidney disease progression in adults with advanced chronic kidney disease (estimated glomerular filtration rate [eGFR] between 15-45 mL/min/1.73 m2) using intensive blood pressure control and intensive lipid management with 2X2 factorial design.

DETAILED DESCRIPTION:
The EXploring approaChEs with Lower targets of blood preSsure and lIpid for impOving Renal outcome in advanced Chronic Kidney Disease (EXCELSIOR-CKD) strived to enroll about 642 participants aged ≥19 years with eGFR 15-45 mL/min/1.73 m2, systolic blood pressure (SBP) ≥130 mmHg, and low-density lipoprotein cholesterol (LDL-C) ≥100 mg/dL.

The EXCELSIOR-CKD study is a 2X2 factorial design with factors consisting of: intensive versus standard SBP control (120 vs 140 mmHg), and intensive versus standard LDL-C control (70 vs 100 mg/dL).

The primary hypothesis was that kidney disease progression event rates would be lower in the intensive arms. Participants would be recruited at 13 clinics over approximately a 2-year period, and are planned to be followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of all of followings

  1. At least 19 years old
  2. Evidence of CKD defined at least 3 months before and at the time of screening visit with CKD-EPI eGFR ≥15 to <45 mL/min/1.73 m2
  3. SBP of

     * 130-180 mmHg on 0 or 1 medication
     * 130-170 mmHg on upto 2 medications
     * 130-160 mmHg on more than 3 medications
  4. LDL-C ≥100 mg/dL

Exclusion Criteria:

* Any of followings

  1. Resistant hypertension or poorly controlled hypertension

     * Failure to achieve SBP of <140 mmHg despite using 4 or more antihypertensive medications including diuretics
  2. Known secondary cause of hypertension
  3. History of renal devervation procedure
  4. Glomerulonephritis requiring immunosuppresive agents
  5. Autosomal dominant polycystic kidney disease receiving tolvaptan
  6. CKD-EPI < 15 mL/min/1.73 m2 or receiving kidney replacement therapy
  7. Familial hypercholesterolemia
  8. Cardiovascular event or precedure (as defined as myocardial infarction, unstable angina, coronary revascularization, or stroke) within last 3 months or planning to cardiovascular procedure upcoming 3 months at the time of screening visit
  9. Symptomatic heart failure within 6 months of left ventricular ejection fraction <45%
  10. A medical condition likely to limit survival to less thant 3 years
  11. Diagnosis of malignancy within the last 5 years or undergoing chemotherepy or radiotherapy
  12. Any organ transplant
  13. Advanced cirrhosis (Child-Pugh class B or C) or abnormal liver function test (alanine transaminase or aspartate transaminase ≥1.5 X upper normal limit)
  14. Evidence of active inflammatory muscle disease (polymyositis or dermatomyositis) or creatine kinase elevation (≥3 X upper normal limit)
  15. History of adverse reaction to HMG-CoA reductase inhibitors or ezetimibe
  16. Using any drugs as followings:

      * Nicotinic acid
      * Macrolide antibiotics
      * Systemic imidazole or triazole antifungal agent
      * Protease inhibitor
      * Nefazodone
      * Immunosuppressive agents (glucocorticoid [equivalent to prednisone 10 mg/day over 4 weeks], cyclosporin, mycofenolate, azathioprine, methotrexate, cyclophosphamide, or rituximab)
  17. Pregnancy or trying to become pregnant
  18. Diabetes mellitus, type I
  19. Diabetes mellitus, type II with HbA1c ≥10.0%

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Renal composite outcome | up to 3 years
  Renal composite outcome would be defined as one of followings:
  1. A sustained decline in eGFR of 40%,
  2. Initiation of kidney replacement therapy (dialysis or kidney transplantation),
  3. A sustained eGFR <10 mL/min/1.73 m2, or
  4. Death from renal causes

SECONDARY OUTCOMES:
Individual components of renal composite outcome | up to 3 years
  1. A sustained decline in eGFR of 40%
  2. Initiation of kidney replacement therapy (dialysis or kidney transplantation),
  3. A sustained eGFR <10 mL/min/1.73 m2
  4. Death from renal causes
  5. Rate of change of eGFR during chronic phase I (12 week to 3 year)
  6. Rate of change of eGFR during chronic phase II (24 week to 3 year)
  7. Rate of change of eGFR during study period (0 week to 3 year)
  8. Cardiovascular composite outcome (defined as one of followings):
     1. Death from cardiovascular causes,
     2. Non-fatal myocardial infarction,
     3. Non-fatal stroke (ischemic or hemorrhagic),
     4. Hospitalization for heart failure, or
     5. Revascularization (coronary, carotid, or peripheral artery)
eGFR slopes | up to 3 years
  1. A sustained decline in eGFR of 40%
  2. Initiation of kidney replacement therapy (dialysis or kidney transplantation),
  3. A sustained eGFR <10 mL/min/1.73 m2
  4. Death from renal causes
  5. Rate of change of eGFR during chronic phase I (12 week to 3 year)
  6. Rate of change of eGFR during chronic phase II (24 week to 3 year)
  7. Rate of change of eGFR during study period (0 week to 3 year)
  8. Cardiovascular composite outcome (defined as one of followings):
     1. Death from cardiovascular causes,
     2. Non-fatal myocardial infarction,
     3. Non-fatal stroke (ischemic or hemorrhagic),
     4. Hospitalization for heart failure, or
     5. Revascularization (coronary, carotid, or peripheral artery)
Cardiovascular composite outcome | up to 3 years
  1. A sustained decline in eGFR of 40%
  2. Initiation of kidney replacement therapy (dialysis or kidney transplantation),
  3. A sustained eGFR <10 mL/min/1.73 m2
  4. Death from renal causes
  5. Rate of change of eGFR during chronic phase I (12 week to 3 year)
  6. Rate of change of eGFR during chronic phase II (24 week to 3 year)
  7. Rate of change of eGFR during study period (0 week to 3 year)
  8. Cardiovascular composite outcome (defined as one of followings):
     1. Death from cardiovascular causes,
     2. Non-fatal myocardial infarction,
     3. Non-fatal stroke (ischemic or hemorrhagic),
     4. Hospitalization for heart failure, or
     5. Revascularization (coronary, carotid, or peripheral artery)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park CH, Kim HW, Park JT, Chang TI, Yoo TH, Oh KH, Anderson AH, Yang W, Cohen JB, Rahman M, Kang SW, Han SH; on the behalf of CRIC Study and KNOW-CKD Investigators. BP and Kidney Disease Progression in Advanced CKD: Findings from the Chronic Renal Insufficiency Cohort and KoreaN Cohort Study for Outcome in Patients with CKD Studies. Clin J Am Soc Nephrol. 2025 Jun 6;20(9):1179-1189. doi: 10.2215/CJN.0000000760. PMID 40478754